CLINICAL TRIAL: NCT01988389
Title: Effect of Apples Consumption on Blood Lipid Levels,Vascular Function and Gut Health in Moderate Hypercholesterolemic Subjects
Brief Title: Effect of Apples on cardioVascular Risk And Gut Health
Acronym: AVAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Fondazione Edmund Mach di San Michele all'Adige (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 13/22; University of Reading
Record Dates: First submitted 2013-10-10; First posted 2013-11-20 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Mild Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- whole apples (Experimental): Subjects are asked to consume 2 apples a day for 8 weeks in addition to their habitual diet
  Interventions: Dietary Supplement: whole apples (WA)
- apple juice squash (Other): Subjects are asked to consume 100 ml of apple juice squash (recommended dilution with water up to 500 ml) for 8 weeks in addition to their habitual diet. The apple juice is used as a sugar matched control.
  Interventions: Dietary Supplement: apple juice (AJ)

INTERVENTIONS:
Dietary Supplement: whole apples (WA)
  Arms: whole apples
Dietary Supplement: apple juice (AJ)
  Arms: apple juice squash

SUMMARY:
There is now considerable scientific evidence that a diet rich in fruits and vegetables could improve human health. Apples are among the most frequently consumed fruits in the world. Epidemiological studies have linked frequent apple consumption with several health benefits including a reduced risk of cardiovascular disease. Apples are an important source of polyphenols and fiber and their beneficial effects could be attributed to this content; however, their impact on our health is not clear. Although, there are some studies that have reported cholesterol lowering effects the results are inconsistent. Furthermore, few studies have explored the impact on vascular function and gut microbiota. The objective of the current study is to assess whether a regular apple consumption, reduces total cholesterol levels, improves vascular function and gut microbiota profile in mildly hypercholesterolemic subjects compared with a control, sugar matched commercial clear apple juice squash.

ELIGIBILITY:
Inclusion Criteria:

* Mildly hypercholesterolemic: TC>5.2 and <7.9 mmol/L
* BMI: 20-35
* Age: 23-69
* Normal liver and kidney function

Exclusion Criteria:

* Drug treatment for hyperlipidaemia, hypertension, inflammation and hypercoagulation.
* Vegetarians.
* Smoking.
* History of alcohol misuse.
* History of food allergy (e.g. apples, sulphites).
* Taking antibiotics for the previous 3 months.
* Taking phytochemical, antioxidant, fish oil supplements, or prebiotic/probiotic preparations unless willing to stop for the study period and after a 4 week wash out period (8 weeks for fish oil).
* Females who are pregnant, lactating, or if of reproductive age and not using a reliable form of contraception (including abstinence).
* Medical history of cardiovascular disease including coronary heart disease (angina and heart attack) and stroke (in the past 12 months).
* Family history of cardiovascular disease (their father or brother was under 55 or their mother or sister was under 65 when they were diagnosed with cardiovascular disease).
* Diabetes mellitus.
* Kidney, liver, pancreas or gastrointestinal diseases.
* Hematologic disorders (i.e. anaemia; men:haemoglobin<13.8g/dl (8.56mmol/L) and women<12.1 g/dl (5.51mmol/L)).
* Planning a weight reducing regime.
* Parallel participation in another dietary intervention study.

Ages: 23 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in blood lipid levels | Baseline and assessment at 8 weeks for each intervention arm including a 4 week wash out period.

SECONDARY OUTCOMES:
Evaluation of endothelial function by using laser doppler iontophoresis (LDI) | Baseline and assessment at 8 weeks for each intervention arm.
Changes in vascular stiffness by pulse wave analysis (PWA) | Baseline and assessment at 8 weeks for each intervention arm
Changes in faecal bacterial population | Baseline and assessment at 8 weeks for each intervention arm
Ambulatory blood pressure | Baseline and assessment at 8 weeks for each intervention arm
  Blood pressure will be recorded for 30 minutes at baseline and at 8 weeks for each intervention arm
Changes in inflammatory, endothelial function and oxidative stress markers | Baseline and assessment at 8 weeks for each intervention arm
Changes in insulin resistance and gut hormones | Baseline and assessment at 8 weeks for each intervention arm
Metabolomic analysis for the determination of the low molecular weight metabolite profiles in the biological fluids (blood, urine and faecal sample). | Baseline and assessment at 8 weeks for each intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, BSc, PhD, RNutr, Principal Investigator — University of Reading; Kieran Tuohy, Dr, Principal Investigator — FEM-IASMA Research and Innovation centre
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Koutsos A, Riccadonna S, Ulaszewska MM, Franceschi P, Trost K, Galvin A, Braune T, Fava F, Perenzoni D, Mattivi F, Tuohy KM, Lovegrove JA. Two apples a day lower serum cholesterol and improve cardiometabolic biomarkers in mildly hypercholesterolemic adults: a randomized, controlled, crossover trial. Am J Clin Nutr. 2020 Feb 1;111(2):307-318. doi: 10.1093/ajcn/nqz282. PMID 31840162